CLINICAL TRIAL: NCT00617032
Title: A Phase 1 Dose Escalation Study of Intra-Articular Administration of tgAAC94, a Recombinant Adeno-Associated Vector Containing the TNFR:Fc Fusion Gene, in Inflammatory Arthritis
Brief Title: Phase 1 Dose Escalation Study of Intra-Articular Administration of tgAAC94
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Targeted Genetics Corporation (Industry)
Responsible Party: Rae Saltzstein, Senior Director Quality and Regulatory Affairs, Targeted Genetics Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13E04; RAC Protocol # 0307-588; HPB 0088676
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 1x10^10 DRP/mL tgAAC94
  Interventions: Genetic: tgAAC94 gene therapy vector
- 2 (Active Comparator): 1x10^11 DRP/mL tgAAC94
  Interventions: Genetic: tgAAC94 gene therapy vector
- 3 (Placebo Comparator): Single dose tgAAC94 placebo
  Interventions: Genetic: tgAAC94 placebo

INTERVENTIONS:
Genetic: tgAAC94 gene therapy vector — Single Dose 1x10^10 DNase resistant particles (DRP) / mL joint volume
  Arms: 1
Genetic: tgAAC94 gene therapy vector — Single dose 1x10^11 DNase resistant particles (DRP) / mL joint volume
  Arms: 2
Genetic: tgAAC94 placebo — Single dose
  Arms: 3

SUMMARY:
Study 1304 is a Phase I dose escalation study conducted in adults with persistent moderate (grade 2) or severe (grade 3) swelling due to inflammatory arthritis (rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis) in at least one peripheral joint eligible for injection. Disease must not be severe enough to warrant use of a TNF-alpha antagonist in the next three months.

Current use of TNF-alpha antagonists is not permitted. Subjects with rheumatoid arthritis must have had an adequate trial of at least one disease-modifying antirheumatic drug (DMARD) prior to screening.

The primary objective is to evaluate the safety of intra-articular administration of tgAAC94.

DETAILED DESCRIPTION:
tgAAC94 is a recombinant adeno-associated virus serotype 2 (AAV2) vector genetically engineered to contain the cDNA for a human tumor necrosis factor receptor (TNFR)-immunoglobulin (IgG1) Fc fusion (TNFR:Fc) gene. The DNA sequence of TNFR:Fc in tgAAC94 codes for a protein sequence identical to etanercept (Enbrel). TNF-alpha has been strongly implicated as a major participant in the inflammatory cascade that leads to joint damage and destruction in diseases such as rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS).

Intra-articular delivery of the TNFR:Fc gene (tgAAC94) should result in expression of the secreted protein in the joint space and provide local high concentrations of soluble TNFR:Fc for an extended period of time without requiring frequent administration. Thus, this proposed therapy would be useful in those inflammatory arthritis patients who have a persistently problematic joint despite the use of systemic TNF-alpha blockade or who have a limited number of arthritic joints.

Extensive preclinical studies using rAAV2 containing several different transgenes in a variety of animal models have shown efficient and persistent gene transfer and expression with minimal toxicity. The parent virus (wild-type AAV2) is a naturally occurring, non-replicating virus that depends on a helper virus, such as adenovirus, for replication. The recombinant AAV2 vector is unable to replicate in target host cells because it lacks the AAV genes, whose protein products are also required in trans, for replication and packaging of progeny virus. Extensive epidemiological studies have found AAV2 to be non-pathogenic.

Although there is no cure for inflammatory arthritis, treatment has been revolutionized by the advent of anti-TNF-alpha therapies. These include etanercept (Enbrel), infliximab (Remicade) and adalimumab (Humira), which consist of soluble TNF receptors, chimeric human-mouse anti-TNF-alpha monoclonal antibodies and fully human anti-TNF-alpha monoclonal antibodies, respectively. Clinical studies have shown these products to improve the signs and symptoms, inhibit the structural damage, and impact functional outcomes in patients with inflammatory arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis, diagnosed according to published criteria
* Persistent moderate (grade 2) or sever (grade 3) swelling due to inflammatory arthritis in at least one peripheral joint eligible for injection
* For subjects with rheumatoid arthritis, an adequate trial of at least one disease-modifying antirheumatic drug (DMARD) prior to screening
* For subjects currently on DMARD(s), a stable regimen for inflammatory arthritis for the previous three months, with no changes in doses in the four weeks prior to screening
* Age greater than 18 years
* Be willing to practice effective birth control measures during the study, if of reproductive ability
* Able to give written informed consent

Exclusion Criteria:

* Current use of a TNF-alpha antagonist
* Disease severe enough to warrant use of a systemic TNF-alpha antagonist in the next three months
* Discontinuation of TNF-alpha antagonists in the past because of safety concerns
* Current use of anakinra
* Poor functional status, defined as being bed-bound or wheelchair-bound
* Corticosteriod therapy at doses higher than the equivalent of 10 mg prednisone per day
* Any of the following laboratory values: Hemoglobin <8.5 gm/dL, white blood cell count <3500 per mm^3, platelet <100 K/microL, creatinine >2 mg/dL, bilirubin >2 mg/dL, AST or ALT >2 times the upper limit of normal, or abnormal coagulation profiles
* Known HIV infection, known hepatitis C infection, or known positive serologic test for hepatitis B surface antigen
* Positive PPD, unless previously treated with appropriate prophylaxis
* Pregnancy or lactation, either at the time of screening or planned in the next six months
* Inflammatory bowel disease, such as Crohn's disease or ulcerative colitis
* Serious medical disease, such as sever liver or kidney disease, uncompensated congestive heart failure, myocardial infarction within six months, unstable angina, uncontrolled hypertension, severe pulmonary disease or active asthma, demyelinating neurological disease, history of cancer (other than cutaneous basal and squamous cell carcinoma) with less than five years documentation of a disease free state, insulin-dependent diabetes, recurrent opportunistic infections or other concurrent medical condition that, in the opinion of the investigator, would make the subject unsuitable for the study
* Unlikely to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | From study drug administration through final study visit
Severe or very severe adverse events | From study drug administration through final study visit
Study drug-related adverse events | From study drug administration through final study visit

SECONDARY OUTCOMES:
Change in tenderness and swelling of injected joint | Days 3 and 7 and Weeks 2, 4, 8, and 12
Change in tenderness and swelling of non-injected joints | Weeks 2, 4, and 12
Reduction in disease activity, as measured by American College of Rheumatology (ACR) criteria and Disease Activity Score (DAS) | Weeks 2, 4, and 12
Joint fluid measures (cell count and differential, total protein and TNFR:Fc protein) | Weeks 4 and 12
TNFR:Fc protein levels in serum | Day 7 and Weeks 2, 4, 8, and 12
Serum neutralizing antibodies to AAV2 | Weeks 4 and 12
Presence of tgAAC94 in peripheral blood mononuclear cells (PBMCs) | Day 3 and Weeks 2 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Study Director — Targeted Genetics Corporation
Locations (7):
- United States (3):
  - UCLA Division of Rheumatology, Los Angeles, California
  - Denver Arthritis Research Center, Denver, Colorado
  - Swedish Rheumoatology Research, Seattle, Washington
- Canada (4):
  - Arthritis Research Centre of Canada, Vancouver, British Columbia
  - Arthritis Centre Clinical Research Unit UofManitoba, Winnipeg, Manitoba
  - Mt Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario